CLINICAL TRIAL: NCT05058196
Title: Choice And Real Experience of Therapeutic deEscalation in Women Over 65 Year With Breast Cancer (CARTE)
Brief Title: Patient's Choice in the Reduction of Their Treatment in Women Over 65 Year With Breast Cancer
Acronym: CARTE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0107/1903
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Therapeutic de-escalation; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Whole breast radiotherapy after surgery (Other): WBRT will be delivered at 50 Grays (2 Grays x 25 fractions), 5 days/week for 5 weeks after breast surgery
  Interventions: Radiation: Whole breast radiotherapy
- Intra Operative Radiotherapy (Other): IORT will be delivered at a single dose of 20 grays to the tumor bed during breast surgery
  Interventions: Radiation: Intra Operative Radiotherapy
- no radiotherapy (No Intervention): No radiotherapy will be administrated to the patients during or after breast surgery

INTERVENTIONS:
Radiation: Whole breast radiotherapy — Whole breast radiotherapy after surgery
  Arms: Whole breast radiotherapy after surgery
Radiation: Intra Operative Radiotherapy — Intra Operative Radiotherapy
  Arms: Intra Operative Radiotherapy

SUMMARY:
Standard treatment for women with early breast cancer (HR+, HER2-, T1N0) consists of the removal of the tumor from the breast by surgery with or without chemotherapy, followed by a whole-breast radiation therapy (usually one radiation treatment a day, five days a week, for 3 to 6 weeks)

In some cases, for elderly patients older than 65 years with other associated pathologies, therapeutic de-escalation might be proposed in order to reduce the radiation doses received. Two options can be considered:

* Intraoperative radiotherapy: radiation is delivered in a single dose directly to the tumor bed during the surgery.
* Radiotherapy omission

These three treatment options (whole-breast radiation therapy, Intraoperative radiotherapy or -Radiotherapy omission) have advantages and disadvantages. Intraoperative radiotherapy allows a targeted treatment and avoids several weeks of daily radiation. Radiotherapy omission prevents acute or late toxicities of the radiotherapy, as well as the constraints of daily travel over a period of 3 to 6 weeks.

The aim of this trial is to offer patients aged 65 and over with early breast cancer, after surgery, these three treatment options and to study the choice and experience of treatment by patients. This study will assess the reasons that prompted patients to choose one of the three treatment options, the impact of medical and personal characteristics on this choice and the experience of therapeutic de-escalation as well as its effects, in particular on the course of care.

This assessment will be carried out with self-administered questionnaires before and after the choice of treatment.

In addition, to standardize the information given to patients in order to support them in their treatment choice and promote patient involvement in treatment decision-making, an encounter decision aid will be available for the patients. This encounter will detail the advantages and disadvantages of the three treatment options and will help in discussions with the physicians to determine the best choice of treatment.

DETAILED DESCRIPTION:
Current demographic trends lead to an increasing number of breast cancers among 70+ women. In this population, adjuvant whole-breast radiation therapy (WBRT) after breast conserving surgery has proven its advantage on local control, but does not improve survival. Some experts are thus advocating WBRT omission.

In this context of limited life expectancy and of frequent comorbidities, therapeutic de-escalation (DE) might be proposed. Two options of de-escalation have been considered: (1) omission of adjuvant breast irradiation and (2) limiting the breast irradiated volume through a single-dose targeted intraoperative radiotherapy (IORT). As each of the three options (standard WBRT, IORT or no irradiation at all) has significant harms and benefits, treatment decision-making should not rely on the physician's opinion only.

A recent study has shown that in this context older women desire information and have more agency and input in the decision-making process than prior literature would suggest. The impact of therapeutic de-escalation on objective indicators and on patient reported outcomes must be investigated in current clinical practice, as uncertainties and doubt are likely to affect the decision-making process. When there is no definitive evidence to favour a treatment decision, assessing the patients' values and preferences appear to be of great relevance and value. Thus, the impact of therapeutic de-escalation on objective indicators and on patient reported outcomes (PROs) and experience (PRE) must be investigated, as uncertainty is likely to affect the decision-making process. We therefore propose to study the women's choice and experience of de-escalation of radiotherapy.

An encounter decision aid will be used to standardize the information provided about the three options and their outcomes. A prospective multicentre study using self-administered questionnaires before and after treatment decision making will then examine:

* the patient's choice and the impact of medical and patients' characteristics on this choice,
* the reason for the therapeutic choice from the patient's point of view,
* the experience of DE (patient-reported outcomes), and its medical effects (including care trajectories).

This study will document the rate and reasons of DE choice among French elderly early breast cancer patients. The results should facilitate the physician's reasoning at the time of treatment decision, and will also help patients (and their relatives) become better informed of the potential consequences of their choices. Developing a patient decision aid might also promote higher quality choices and shared decision-making in this context.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent form prior to any study specific procedures; when the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor can confirm in writing the patient's consent
2. Women ≥65 years of age
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤2
4. Clinical stage I, newly diagnosed breast cancer; invasive unifocal HR+ HER2- T1N0 tumour, not lobular, without extensive intraductal component (EIC) (<25% EIC on biopsy), without embolism on biopsy
5. Eligible to surgery
6. Eligible for both WBRT or IORT
7. Chemotherapy treatment is possible if needed
8. Able to respond to self-report questionnaires in French
9. Affiliated to Social security System

Exclusion Criteria:

1. Patient with recurrent breast cancer or inflammatory breast carcinoma
2. Absolute contra-indication to whole-breast irradiation as determined by the referring physician
3. Patient unable to comply with study obligations for geographic, social, or physical reasons, or who is unable to understand the purpose and procedures of the study
4. Patient enrolled in another therapeutic trial. Observational cohorts are accepted if the collection of data does not interfere with the current trial
5. Person deprived of their liberty or under protective custody or guardianship.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Patient's choice when de-escalation is proposed between whole breast radiotherapy (WBRT), Intra Operative Radiotherapy (IORT) or no radiotherapy (RT). | At baseline
  Assess the rate for each strategy of treatment chosen (WBRT, IORT or no RT) (decision made) by the patient.

SECONDARY OUTCOMES:
Final treatment received (WBRT, IORT or no RT) | 6 weeks maximum (two weeks after surgery)
  Collection of final treatment (WBRT, IORT or no RT) to check for potential changes after the decision was made
Reason for the therapeutic choice from the patient's point of view | 6 weeks maximum (two weeks after surgery)
  The patients must indicate the level of importance of the delivered information to decide their treatment strategy option by assigning a score from 0 to 10 (ie, duration of the surgery, number of radiotherapy sessions, need for additional medical examinations ...)
Encounter decision aid (EDA) rate of use | At baseline
  This encounter decision aid has been developed in collaboration with patients, radiation oncologists, communication specialists, and the US research team who developed the first EDAs. The developed EDA presents the main similarities and differences between the 3 treatment options using the main reasons to choose or decline therapeutic de-escalation elicited by the preliminary qualitative study and by previous literature on patients' preferences and information needs.
Geriatric Core Dataset (G-CODE) | At baseline
  The G-CODE is a minimum set of geriatric data to be collected in cancer trials. It was developed after a Delphi consensus method with international agreement. The G-CODE has ten tools/items and a median completion time of 9 min. It allows for a minimal geriatric description of the older cancer population and standardization of geriatric data, enabling comparison across trials. The items within the G-CODE are the following: (1) social assessment: living alone or support requested to stay at home; (2) functional autonomy: Activities of Daily Living (ADL) questionnaire and short instrumental ADL questionnaire; (3) mobility: Timed Up and Go test; (4) nutrition: weight loss during the past 6 months and body mass index; (5) cognition: Mini-Cog test; (6) mood: mini- Geriatric Depression Scale and (7) comorbidity: updated Charlson Comorbidity Index. The total scale range 0-62. High score indicate better condition.
Single Item Literacy Screener (SILS) | At baseline
  The Single Item Literacy Screener (SILS) is a single item instrument designed to identify patients who need help with reading health-related information. The instrument asks one question "How often do you need to have someone help you when you read instructions, pamphlets, or other written material from your doctor or pharmacy?" with possible responses ranging from "1" (never) to "5" (always). The authors identified the cut-off point as "2" in order to capture all patients potentially in need of assistance.
Control Preferences Scale (CPS) | At baseline
  The Control Preferences Scale (CPS) was developed to measure a construct that emerged from a grounded theory of how treatment decisions are made among people with life-threatening illnesses. The control preferences construct is defined as "the degree of control an individual wants to assume when decisions are being made about medical treatment." The CPS consists of five cards that each portrays a different role in treatment decision-making using a statement and a cartoon. These roles range from the individual making the treatment decisions, through the individual making the decisions jointly with the physician, to the physician making the decisions. The CPS involves subjects in making a series of paired comparisons to provide their total preference order over the five cards. These preference orders are analyzed using unfolding theory to determine the distribution of preferences in different populations and the effect of covariates on consumer preferences.
Fear of Cancer Recurrence-Short form (FCRI-SF) | 6 weeks (two weeks after surgery), 7 and 25 months
  The nine-item Fear of Cancer Recurrence Inventory is a short form of the FCRI (nine-item FCRI) and corresponds to the severity subscale of the FCRI (42 items). The nine-item FCRI evaluates the presence and severity of intrusive thoughts associated with FCR. Each item is rated on a Likert scale ranging from 0 ("not at all" or "never") to 4 ("a great deal' or "all the time")
CollaboRATE survey | 6 weeks (two weeks after surgery), 7 and 25 months
  CollaboRATE is a brief patient survey focused on shared decision making. The CollaboRATE questions are as follows: (i) How much effort was made to help you understand your health issues? (ii) How much effort was made to listen to what matters most to you about your health issues? (iii) How much effort was made to include what matters most to you in choosing what to do next? CollaboRATE survey data included responses to the three CollaboRATE questions, each on a 0-9 scale, along with each respondent's age, gender and clinician
VICAN survey | 6 weeks (two weeks after surgery), 7 and 25 months
  VICAN is a French national survey on life conditions of cancers survivors. In particular, the objectives are to study the labour market outcomes, the effect of cancer on an individual's employability, the psychosocial conditions impact (ie, lifestyle behaviours, perceived discrimination, family and social support) and to evaluate the physical, psychological and social needs.
Decisional Conflict Scale (DCS) | 6 weeks (two weeks after surgery), 7 and 25 months
  The Decisional Conflict Scale (DCS) is a self-administered questionnaire that can be used to 1) diagnose a patient's decisional conflict; 2) identify the patient's decision support needs (knowledge, values clarification, support); 3) determine the quality of the decision process; and 4) evaluate the impact of decision support interventions. The DCS comprises 16 items grouped into five sub-scales: certainty, information, clarification of values, support or pressure from others, and the respondent's perception of the quality of the decision process. Each item is measured on a 5-point Likert scale (0 = strongly agree to 4 = strongly disagree). The patient's score is obtained by adding the scores (0-4) for the 16 items, dividing the sum by 16 and then multiplying it by 25
Quality of life questionnaire - Core 30 (QLQ-C30) | 6 weeks (two weeks after surgery), 7 and 25 months
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life Questionnaire - Breast cancer module (QLQ-BR23) | 6 weeks (two weeks after surgery), 7 and 25 months
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30. The QLQ-BR23 contains 23 items incorporating five multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning. In addition, single items assess sexual enjoyment, hair loss and future perspective. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. For all items but sexual functioning and sexual enjoyment, higher scores indicate more severe symptoms.
Quality of Life Questionnaire - Elderly cancer patients module (QLQ-ELD14 ) | 6 weeks (two weeks after surgery), 7 and 25 months
  The EORTC QLQ EDL14 is a self-reporting specific questionnaire developed to assess the quality of life of elderly cancer patients. It addresses generic issues affecting older people with cancer, not covered by the QLQ-C30 or site-specific modules, and can be used in clinical studies that include older patients, regardless of tumour site of health-related quality of life elderly patients with cancer.
  The questionnaire contains 14 items incorporating five scales to assess mobility, worries about others, future worries, maintaining purpose, and illness burden. In addition, two single items assess joint stiffness and family support. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. High scores indicate poor mobility, good family support, much worry about the future, good maintenance of autonomy and purpose, and high burden of illness.
Decision Regret Scale | 6 weeks (two weeks after surgery), 7 and 25 months
  The Decision Regret Scale is a 5-item Likert-type measure written to assess regret or remorse following a medical decision. Patients respond to the items after reading the prompt: "Please think about the decision you made about [chosen health care decision] after talking to your [doctor, surgeon, nurse, health professional, etc.]." Scores range from of 0 to 100. High scale scores represent higher regret over a health care decision.
Anxiety Level Scale (ALS) | 6 weeks (two weeks after surgery), 7 and 25 months
  Anxiety level Scale (ALS) is 1-item tool developed to measure patient' anxiety. The score range is from 1 to 5. A high scale score represents a higher response level (The score 5 is the level for extremely anxious).
Incidence of Treatment-Emergent Adverse Events | 6 weeks (two weeks after surgery), 7 and 25 months
  The safety will be evaluated by toxicities assessed using the the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) which is widely accepted in the community of oncology research as the leading rating scale for adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Julien MANCINI, MD, PhD, Principal Investigator — Equipe "Cancers Biomédecine & Société" (CANBIOS) UMR1252 SESSTIM, Institut Paoli Calmettes; Agnès TALLET, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.